CLINICAL TRIAL: NCT01623479
Title: An Observational Study of Patients Treated With Bimatoprost 0.03% (Latisse®) for Hypotrichosis of the Eyelashes
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: GMA-LTS-10-001; CED2009 (Other: Allergan)
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2012-09-19 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Eyelash Hypotrichosis
MeSH Terms: interventions — Bimatoprost

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypotrichosis of the Eyelashes: Subjects with hypotrichosis of the eyelashes using bimatoprost 0.03% (Latisse®) as prescribed by physician for at least 12 months
  Interventions: Drug: bimatoprost 0.03%

INTERVENTIONS:
Drug: bimatoprost 0.03% — Subjects with hypotrichosis of the eyelashes using bimatoprost 0.03% (Latisse®) as prescribed by physician for at least 12 months
  Other Names: Latisse®

SUMMARY:
This is an observational study of patients treated with bimatoprost 0.03% (Latisse®) for at least 12 months for hypotrichosis of the eyelashes.

ELIGIBILITY:
Inclusion Criteria:

* Hypotrichosis of the eyelashes
* Using bimatoprost ophthalmic solution 0.03% (Latisse®) for at least 12 months

Exclusion Criteria:

* Use of any over-the-counter medication(s) for eyelash growth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with hypotrichosis of the eyelashes
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2010-11-19 (Actual); Primary Completion 2011-09-01 (Actual); Study Completion 2011-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Santa Ana, California, United States

REFERENCES:
- [Background] Yoelin SG, Fagien S, Cox SE, Davis PG, Campo A, Caulkins CA, Gallagher CJ. A retrospective review and observational study of outcomes and safety of bimatoprost ophthalmic solution 0.03% for treating eyelash hypotrichosis. Dermatol Surg. 2014 Oct;40(10):1118-24. doi: 10.1097/01.DSS.0000452658.83001.d9. PMID 25229783

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hypotrichosis of the Eyelashes
Started | 585
Completed | 585
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Hypotrichosis of the Eyelashes
Number analyzed (Participants) | 585
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.54 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 580
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Satisfied With Latisse®
Description: Overall subject satisfaction with Latisse® was assessed on a 5-point scale (Very Satisfied, Satisfied, Neutral, Unsatisfied, and Very Unsatisfied). The percentage of subjects satisfied and very satisfied is reported.
Time Frame: Day 1
Population: Subjects with all study data
Measure: Number; unit: Percentage of Subjects
Arm/Group | Hypotrichosis of the Eyelashes
Number analyzed (Participants) | 585
Percentage of Subjects | 92.48

2. Secondary Outcome: Number of Applications of Latisse® Per Week
Description: Number of applications of Latisse® per week as reported by the subjects.
Time Frame: Day 1
Population: Subjects with all study data
Measure: Mean (Standard Deviation); unit: Number of Applications
Arm/Group | Hypotrichosis of the Eyelashes
Number analyzed (Participants) | 585
Number of Applications | 6.69 (1.13)

3. Secondary Outcome: Percentage of Subjects Satisfied Wtih Their Eyelashes
Description: Overall subject satisfaction with their eyelashes was assessed on a 5-point scale (Very Satisfied, Satisfied, Neutral, Unsatisfied, and Very Unsatisfied). The percentage of subjects satisfied and very satisfied is reported.
Time Frame: Day 1
Population: Subjects with all study data
Measure: Number; unit: Percentage of Subjects
Arm/Group | Hypotrichosis of the Eyelashes
Number analyzed (Participants) | 585
Percentage of Subjects | 79.81

ADVERSE EVENTS:
Arm/Group | Hypotrichosis of the Eyelashes
Serious Adverse Events (participants affected / at risk) | 0/585
Other Adverse Events (participants affected / at risk) | 155/585
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Hypotrichosis of the Eyelashes (N=585)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 51
Erythema of the Eyelid (Eye disorders) | 35
Eye Pruritus (Eye disorders) | 36
Ocular Irritation (Eye disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.